CLINICAL TRIAL: NCT01871831
Title: Prüfung Von Blutzuckermesssystemen - Bewertung Der Sauerstoffabhängigkeit
Brief Title: Assessment of Blood Glucose Monitoring Systems - Evaluation of Oxygen Dependency
Acronym: IDT-1326-IU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut für Diabetes-Technologie Forschungs- und Entwicklungsgesellschaft mbH an der Universität Ulm (Other)
Collaborators: Roche Diagnostics GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: IDT-1326-IU
Record Dates: First submitted 2013-05-29; First posted 2013-06-07 (Estimated); Last update posted 2015-01-14 (Estimated); Status verified 2013-10

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus | interventions — Self-Testing

INTERVENTIONS:
Device: 6 blood glucose monitoring systems for self-testing

SUMMARY:
Systems for blood glucose monitoring with glucose oxidase enzyme reaction on test strips can be affected by the partial pressure of oxygen of the blood sample. In this study, we investigate the influence of different partial pressure of oxygen in blood samples on measurement results. Systems with labelled oxygen-dependency as well as systems without labelled oxygen-dependency are evaluated.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* male or female subjects with type 1 or type 2 diabetes or healthy subjects
* signed informed consent form

Exclusion Criteria:

* pregnancy or lactation period
* severe acute illness that, in the opinion of the investigator, might pose additional risk to the subject
* severe chronic illness that, in the opinion of the investigator, might pose additional risk to the subject

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2013-06; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Influence of the blood sample's partial pressure on blood glucose measurement results | For each sample, preparation and measurment procedure have an expected duration of about 2 hours

CONTACTS AND LOCATIONS:
Overall Officials: Cornelia Haug, MD, Principal Investigator — Institut für Diabetes-Technologie Forschungs- und Entwicklungsgesellschaft an der Universität Ulm
Locations (1):
- Institut für Diabetes-Technologie Forschungs- und Entwicklungsgesellschaft an der Universität Ulm, Ulm, Germany

REFERENCES:
- [Result] Baumstark A, Schmid C, Pleus S, Haug C, Freckmann G. Influence of partial pressure of oxygen in blood samples on measurement performance in glucose-oxidase-based systems for self-monitoring of blood glucose. J Diabetes Sci Technol. 2013 Nov 1;7(6):1513-21. doi: 10.1177/193229681300700611. PMID 24351177
- See also: Related Info — http://www.ncbi.nlm.nih.gov/pubmed/24351177